CLINICAL TRIAL: NCT02357836
Title: Phase 0 Pharmacodynamic Study of the Effects of Itraconazole on Tumor Angiogenesis and the Hedgehog Pathway in Early-stage Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Itraconazole in Non-small Cell Lung Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, David E Gerber, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122014-038
Record Dates: First submitted 2015-01-15; First posted 2015-02-06 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Itraconazole (Other): 600 mg twice daily for 10-14 days
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Once on study, itraconazole will be taken twice daily for a total of 10-14 days. After being on itraconazole for 7-10 days, "Post-treatment" assessments will include a skin biopsy, blood draw for the PK (pharmacokinetics) analyses and the cytokine panel, and also MRI evaluations (anticipated to last 45-50 minutes). Toxicity assessments and laboratory checks will also be conducted during that time. Following these assessments, itraconazole will be continued until the day of surgery. At the time of surgical resection, a tissue sample (with adjacent normal tissue as per standard resection technique) will be obtained to complete the analysis. Following resection, subjects will be followed per standard post-operative procedure.

SUMMARY:
The purpose of this study is to determine the pharmacodynamics effects of itraconazole in early-stage non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a phase 0 clinical trial. While clinical data including safety will be recorded, the principal outcomes are pharmacodynamic endpoints. Specifically, the investigators seek to identify: (1) effects of itraconazole on tumor angiogenesis, (2) effects of itraconazole on the Hh pathway, (3) biomarker predictors of these effects, (4) the correlation between itraconazole pharmacokinetics and these effects, (5) the correlation between different biomarkers.

Up to 15 eligible patients with previously diagnosed or suspected NSCLC planned for resection will undergo a study-specific core needle biopsy, imaging (dynamic contrast enhanced [DCE]-, diffusion weighted imaging [DWI]-, and arterial spin labeling [ASL] magnetic resonance imaging [MRI]), skin punch biopsy, and collection of peripheral blood. Subjects will then receive itraconazole 600 mg PO daily for 7-10 days, following which they will undergo repeat imaging, skin biopsy, and blood collection. Subsequently they will undergo surgical resection. Due to the safety profile of itraconazole when used as an antifungal agent , all histologic subtypes of NSCLC will be eligible for the trial. The itraconazole dose of 600 mg, higher than an anti-angiogenic dose, has been shown to inhibit the Hedgehog (Hh) pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven NSCLC planned for surgical resection. All NSCLC histologic subtypes are eligible. Alternatively, patients in whom a diagnosis of NSCLC is highly suspected based on history and imaging studies and who are, therefore, scheduled for diagnostic biopsy and/or surgical resection will also be eligible for screening, enrollment, and study treatment if they meet all additional eligibility criteria. In the event that biopsies do not confirm NSCLC, such patients will be removed from study but monitored for any adverse events resulting from study participation.
2. No prior therapy but planned for surgical resection
3. Age ≥ 18 years.
4. ECOG (Eastern Cooperative Oncology Group) 0-2 performance status
5. Adequate organ function as defined below:

   * total bilirubin within normal institutional limits
   * AST (Aspartate Aminotransferase) (SGOT)/ALT (Alanine Aminotransferase) (SPGT) ≤ 2.5 X institutional upper limit of normal
   * creatinine ≤ 2 X institutional upper limit of normal
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   6.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
7. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Subjects may not be receiving any investigational agents that would confound interpretation of study pharmacodynamic endpoints.
2. History of allergic reactions attributed to itraconazole or to compounds of similar chemical or biologic composition to itraconazole.
3. Uncontrolled, concurrent medical illness.
4. Active hepatitis or symptomatic liver disease.
5. History of or current evidence of uncontrolled cardiac ventricular dysfunction (congestive heart failure) or NYHA (New York Heart Association) Class III or IV heart failure.
6. Current use of medications significantly affecting metabolism of itraconazole (certain anti-convulsants, corticosteroids). See 3.5 Drug Interactions in protocol.
7. Current evidence of hyperthyroidism (which would increase metabolism of itraconazole).
8. Pregnant or lactating female or any female trying to get pregnant.
9. Claustrophobia that would interfere with MRI studies anticipated to last 45-50 minutes.
10. Metal implants deemed at risk for migration during MRI studies.
11. CrCl (Creatinine clearance) < 45 mL/min (increased risk of nephrogenic systemic fibrosis [NSF] from MRI Gadolinium contrast).
12. Known allergy to MRI contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Pelosof, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole: 600 mg twice daily for 10-14 days
  Itraconazole: Once on study, itraconazole will be taken twice daily for a total of 10-14 days. After being on itraconazole for 7-10 days, "Post-treatment" assessments will include a skin biopsy, blood draw for the PK analyses and the cytokine panel, and also MRI evaluations (anticipated to last 45-50 minutes). Toxicity assessments and laboratory checks will also be conducted during that time. Following these assessments, itraconazole will be continued until the day of surgery. At the time of surgical resection, a tissue sample (with adjacent normal tissue as per standard resection technique) will be obtained to complete the analysis. Following resection, subjects will be followed per standard post-operative procedure.
Period: Overall Study
Arm/Group | Itraconazole
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Itraconazole
Number analyzed (Participants) | 13
Age, Continuous [Median (Standard Deviation); unit: years] | 64 (0.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 9
  Squamous Cell | 2
  Other | 2
Smoking History [Count of Participants; unit: Participants]
  Former | 10
  Never | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Tumor Tissue Microvessel Density [MVD] From Baseline
Description: Images of DAPI (4',6-Diamidino-2-Phenylindole) , CD31 (cluster of differentiation 31 ), and CD34 (cluster of differentiation 34) were taken from the same field of view and then merged.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Measure: Mean (Standard Deviation); unit: Percent area fraction
Arm/Group | Itraconazole
Number analyzed (Participants) | 13
Percent area fraction | 0.005 (0.045)

2. Secondary Outcome: Change in HIF1α From Baseline
Description: A commercially available kit will be used to measure HIF1α levels.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: We did not collect this data as we did not perform this assay.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in VEGFR2 From Baseline
Description: A commercially available kit will be used to measure VEGFR2 levels.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: We did not collect this data as we did not perform this assay.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Phospho-VEGFR2 From Baseline
Description: A commercially available kit will be used to measure Phospho-VEGFR2 levels.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: We did not collect this data as we did not perform this assay.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

5. Secondary Outcome: Mean Percent Change in Other Plasma Cytokine From Baseline to Post-Treatment
Description: The following plasma cytokines were measured using a commercially available kit.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: The 2 missing cases not included in this analysis here were due to inability to collect the follow-up sample.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Itraconazole
Number analyzed (Participants) | 11
Percent change
  IL-1b | -14.4159 (117.2143)
  IL-1ra | -16.9648 (72.1061)
  IL-2 | -21.5999 (81.7471)
  IL-4 | -5.0114 (36.6851)
  IL-5 | -13.7573 (71.6122)
  IL-6 | -62.5420 (103.4791)
  IL-7 | -21.9919 (64.4562)
  IL-9 | -0.9209 (56.3665)
  IL-10 | 2.9705 (118.2381)
  IL-12 | -30.0689 (99.9174)
  IL-13 | -16.1310 (75.8152)
  IL-15 | -27.7823 (92.4703)
  IL-17 | -24.3512 (82.8199)
  IP-10 | -16.7481 (60.9495)
  MCP-1 | -11.3317 (34.8165)
  MIP-1a | -14.7291 (76.0138)
  MIP-1b | 0.0767 (57.2234)
  RANTES | 5.1468 (128.1372)
  TNF-a | -18.0238 (44.3590)
  IFN-g | -39.7280 (62.7207)
  Eotaxin | 2.8770 (31.7644)
  G-CSF | -4.4567 (30.0457)
  GM-CSF | -45.6701 (60.2840)

6. Secondary Outcome: Mean Percent Change in Angiogenic Cytokines From Baseline
Description: A commercially available kit will be used to measure Angiogenic Cytokines levels.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: The 2 missing cases not included in this analysis here were due to inability to collect the follow-up sample.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Itraconazole
Number analyzed (Participants) | 11
Percent change
  IL-8 | -4.5391 (124.2834)
  PDGF-bb | 7.7116 (209.4990)
  VEGF | -13.5786 (47.4821)
  FGF-b | -35.5341 (65.0768)

7. Secondary Outcome: Changes in Perfusion (Ktrans)
Description: DCE (dynamic contrast enhanced ) MRI is an established technology to assess microvessel density (MVD) and tumor capillary permeability.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: Reasons that enrolled patients did not complete paired research MRI scans included presence of metal implants, inadequate renal function, and patient preference
Measure: Mean (Standard Deviation); unit: min-1
Arm/Group | Itraconazole
Number analyzed (Participants) | 9
min-1 | 0.008 (0.072)

8. Secondary Outcome: Number of Participants With Tumor SMO (Smoothened) Gene Mutations, GLI2 and CCND1 Copy Number, PI3K-mTOR Pathway Activation
Description: phosphatidylinositol-3-kinase (PI3K)/Akt and the mammalian target of rapamycin (PI3K-mTOR pathway )
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: This was initially planned and did not collect data for this and did not assess.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Tumor Tissue GLI1, SHH and PTCH1 Levels From Baseline
Description: This can be measured by analyzing frozen-treated tumor tissue for GLI1 (glioma-associated oncogene ) and PTCH1(patched-1) mRNA (Messenger Ribonucleic Acid) by qPCR.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: The lab tests were not feasible with tumor tissues as they were not enough to conduct these tests.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Skin Biopsy GLI1 Levels From Baseline
Description: We analyzed serial skin biopsies for GLI1 mRNA by qPCR (quantitative polymerase chain reaction).
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: Participant with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: relative units
Arm/Group | Itraconazole
Number analyzed (Participants) | 12
relative units | 0.27347 (0.54713)

11. Secondary Outcome: Change in Skin Biopsy SHH Levels From Baseline
Description: We analyzed serial skin biopsies for SHH (Sonic Hedgehog )levels mRNA by qPCR.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: SHH levels were not measured.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Skin Biopsy PTCH1 Levels From Baseline
Description: We analyzed serial skin biopsies for PTCH1 mRNA by qPCR.
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: Participant with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: relative units
Arm/Group | Itraconazole
Number analyzed (Participants) | 12
relative units | 0.03164 (0.22360)

13. Secondary Outcome: Number of Participants With Tumor Cell Proliferation/Apoptosis
Description: Tumor proliferation and apoptosis will be assessed by tumor Ki67 and cleaved caspase 3 levels
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: This was not feasible with the available tissue samples and hence data not collected.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

14. Secondary Outcome: Itraconazole Levels in Post-treatment Serum
Description: Itraconazole levels assessed by post-treatment serum
Time Frame: Post Treatment (after 7-10 days of itraconazole bid)
Population: The 2 missing cases not included in this analysis here were due to inability to collect the follow-up sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Itraconazole
Number analyzed (Participants) | 11
ng/mL | 1264 (688)

15. Secondary Outcome: Itraconazole Levels in Tumor Tissue
Description: Itraconazole levels assessed by tumor tissue
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: The 4 missing cases not included in this analysis here were due to inability to collect the follow-up sample.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Itraconazole
Number analyzed (Participants) | 9
ng/g | 2585 (1986)

16. Secondary Outcome: Itraconazole Levels in Skin Biopsy
Description: Itraconazole levels assessed by skin biopsy
Time Frame: Baseline and Post Treatment (after 7-10 days of itraconazole bid)
Population: We have not measured itraconazole level in skin biopsy.
Arm/Group | Itraconazole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=13)
Nausea (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 1
Non-Cardiac chest pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02357836/Prot_SAP_000.pdf